CLINICAL TRIAL: NCT01469845
Title: Hypertonic Saline in Acute Bronchiolitis: Randomised Controlled Trial and Economic Evaluation
Brief Title: The SABRE Trial of Hypertonic Saline in Acute Bronchiolitis
Acronym: SABRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCH/1/016; HTA09/91/22 (Other Grant/Funding Number: NHS NIHR HTA)
Record Dates: First submitted 2011-11-09; First posted 2011-11-10 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Acute Bronchiolitis
Keywords: hospital admissions; acute bronchiolitis; under one year old; requiring oxygen therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertonic saline and usual care (Active Comparator)
  Interventions: Device: 3% hypertonic saline
- usual care (oxygen therapy) (Active Comparator)
  Interventions: Device: 3% hypertonic saline

INTERVENTIONS:
Device: 3% hypertonic saline — 4 ml dose to be administered every 6 hours
  Other Names: mucoclear 3%

SUMMARY:
Acute bronchiolitis is a common, distressing illness affecting children. A virus infects the lungs, and then the airways become blocked, leading to difficulties with breathing. It is the most common reason why children are admitted to hospital, with 1-3% of all children admitted to hospital during their first winter, creating enormous strains on NHS services. The majority of those admitted with the condition are under six months of age and the associated stress for parents is considerable. After forty years of research the best treatment we have is supportive care and oxygen.

Recent research suggests that salt water, sprayed as a mist so that the children can breathe it in ('nebulised 3% hypertonic saline') might help children with acute bronchiolitis. Scientists think that the salt water changes the mucus which blocks the airways so that it can be cleared more easily. Three small research studies all suggested that a child's time in hospital could be reduced by a quarter by using this treatment. If this was true, it would be good for children, their families and the children's wards trying to cope with the large numbers admitted with bronchiolitis every year.

To decide whether this treatment should be used throughout the NHS, we need to run a randomised controlled trial of hypertonic saline in a large number of children. The trial will tell us if adding saline to usual care reduces distress in both children and parents, as well as whether it reduces the length of time they stay in hospital. We will then know if the treatment is the best thing for children with bronchiolitis and whether it provides the NHS with good value for money.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy infants under 1 year of age
* Admitted to hospital with a clinical diagnosis of acute bronchiolitis, following the UK definition of an infant with an apparent viral respiratory tract infection associated with airways obstruction manifest by hyperinflation, tachypnoea and subcostal recession with widespread crepitations on auscultation
* Requiring supplemental oxygen therapy on admission

Exclusion Criteria:

* Wheezy bronchitis or asthma - children with an apparent viral respiratory infection and wheeze with no or occasional crepitations
* Previous lower respiratory tract infections
* Risk factors for severe disease [gestation <32 weeks, immunodeficiency, neurological and cardiac conditions, chronic lung disease]
* Subjects where the carer's English is not fluent and translational services are not available
* Requiring admission to high dependency or intensive care units at the time of recruitment

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time to 'fit for discharge' | This was judged to be when the infant was feeding adequately [taking >75% of usual intake] and was in air with a saturation of at least 92% for 6 hours, to reflect clinical practice.
  The primary objective was an analysis, to show if the addition of 3% hypertonic saline to usual care results in significant [25%] reduction in the duration of hospitalisation of infants admitted with acute bronchiolitis. This outcome was measured at 6 hourly intervals, with the first evaluation at time of randomisation.

SECONDARY OUTCOMES:
Actual time to discharge | This was measured from time to randomisation to the discharge time according to routine clinical guidelines.
  The secondary objectives were assessments of the economic impact of such an intervention on both the NHS and parents, as well as quality of life and other health related outcomes assessed 28 days after entry to the study.
Readmission | Within 28 days from randomisation
  The secondary objectives were assessments of the economic impact of such an intervention on both the NHS and parents, as well as quality of life and other health related outcomes assessed 28 days after entry to the study.
health care utilisation | post-discharge and within 28 days from randomisation
  The secondary objectives were assessments of the economic impact of such an intervention on both the NHS and parents, as well as quality of life and other health related outcomes assessed 28 days after entry to the study
duration of respiratory symptoms | post discharge and within 28 days from randomisation
  The secondary objectives were assessments of the economic impact of such an intervention on both the NHS and parents, as well as quality of life and other health related outcomes assessed 28 days after entry to the study
Infant and parental quality of life using the Infant Toddler Quality of Life (ITQoL) questionnaire | 28 days following randomisation.
  The secondary objectives were assessments of the economic impact of such an intervention on both the NHS and parents, as well as quality of life and other health related outcomes assessed 28 days after entry to the study

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Alder Hey Children's NHS Foundation Trust Hospital, Liverpool, Merseyside
  - University Hospital of North Staffordshire, Stoke, North Staffordshire
  - University Hospital of Wales, Cardiff, South Wales
  - Doncaster & Bassetlaw Hospitals NHS Foundation Trust, Doncaster, South Yorkshire
  - Rotherham NHS Foundation Trust, Rotherham, South Yorkshire
  - Sheffield Children's NHS Foundation Trust, Sheffield, South Yorkshire
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire
  - Calderdale and Huddersfield NHS Foundation Trust, Halifax, West Yorkshire
  - Leeds Teaching Hospital NHS Trust, Leeds, West Yorkshire

REFERENCES:
- [Derived] Everard ML, Hind D, Ugonna K, Freeman J, Bradburn M, Dixon S, Maguire C, Cantrill H, Alexander J, Lenney W, McNamara P, Elphick H, Chetcuti PA, Moya EF, Powell C, Garside JP, Chadha LK, Kurian M, Lehal RS, MacFarlane PI, Cooper CL, Cross E. Saline in acute bronchiolitis RCT and economic evaluation: hypertonic saline in acute bronchiolitis - randomised controlled trial and systematic review. Health Technol Assess. 2015 Aug;19(66):1-130. doi: 10.3310/hta19660. PMID 26295732
- [Derived] Everard ML, Hind D, Ugonna K, Freeman J, Bradburn M, Cooper CL, Cross E, Maguire C, Cantrill H, Alexander J, McNamara PS; SABRE Study Team. SABRE: a multicentre randomised control trial of nebulised hypertonic saline in infants hospitalised with acute bronchiolitis. Thorax. 2014 Dec;69(12):1105-12. doi: 10.1136/thoraxjnl-2014-205953. PMID 25389139
- See also: Study specific website — http://www.shef.ac.uk/scharr/sabre